CLINICAL TRIAL: NCT02739269
Title: A Randomised Trial to Compare Antral Follicle Count and Serum Anti-Mullerian Hormone Level for Determination of Gonadotrophin Dosing in In-vitro Fertilisation
Brief Title: Antimullerian Hormone Versus Antral Follicle Count for Determination of Gonadotrophin Dosing in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Hang Wun Raymond Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: UW 12-358
Record Dates: First submitted 2016-04-04; First posted 2016-04-15 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Infertility
Keywords: ovarian response; anti-Mullerian hormone; antral follicle count
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMH group (Active Comparator): Serum AMH measurement
  Interventions: Other: Serum AMH measurement
- AFC group (Sham Comparator): AFC measurement
  Interventions: Other: AFC measurement

INTERVENTIONS:
Other: Serum AMH measurement — Serum AMH is measured one month before the IVF treatment
  Arms: AMH group
Other: AFC measurement — Early follicular phase AFC is measured one month before the IVF treatment
  Arms: AFC group

SUMMARY:
This is a prospective randomized trial to compare the use of AFC and serum AMH as the basis for gonadotrophin dosing in in-vitro fertilization treatment.

The hypothesis is that the use of serum AMH as the criterion for determination of gonadotrophin dosing in IVF treatment results in more optimal ovarian response than AFC.

DETAILED DESCRIPTION:
Patients undergoing the first-time IVF treatment cycle using either conventional insemination technique or intracytoplasmic sperm injection at Queen Mary Hospital will be invited to participate in this study. Participating subjects will be randomized into either (i) AFC or (ii) AMH group, where the gonadotrophin dosing will be determined based on the baseline AFC and serum AMH respectively as assessed one month before the IVF treatment. Randomisation will be performed according to a computer-generated list which will be read by an independent research nurse. That research nurse will assign the initial gonadotrophin dose according to the study protocol.

In the AFC group, starting dose of gonadotrophin will be determined based on serum AMH concentration as follows:

AFC <= 5: 300 IU daily AFC >5 and <=15: 225 IU daily AFC >15: 150 IU daily

In the AMH group, starting dose of gonadotrophin will be determined based on serum AMH concentration as follows:

AMH <= 1.0 ng/ml: 300 IU daily AMH >1.0 and <=3.3 ng/ml: 225 IU daily AMH >3.3 ng/ml: 150 IU daily

The clinician and patient will both be blinded to the randomization throughout the course of treatment. The proportion of subjects having appropriate ovarian response, defined as the number of oocytes retrieved being 6 to 14 inclusive, will be compared between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing the first IVF cycle during the study period.

Exclusion Criteria:

* Body mass index >=30 kg/m2
* Subjects in repeated IVF cycles
* Subjects undergoing IVF treatment using donor oocytes
* Subjects undergoing pre-implantation genetic diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hang Wun Raymond Li, MBBS, FRCOG, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
No such plan at the moment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 women who were undergoing in vitro fertilisation treatment in Queen Mary Hospital, Hong Kong, were recruited.
Groups:
- AMH Group: Serum AMH measurement
  Gonadotrophin dosing was based on serum AMH measured one month before the IVF treatment
- AFC Group: AFC measurement
  Gonadotrophin dosing was based on early follicular phase AFC measured one month before the IVF treatment
Period: Overall Study
Arm/Group | AMH Group | AFC Group
Started | 100 | 100
Completed | 93 | 96
Not Completed | 7 | 4
Not completed — Protocol Violation | 5 | 0
Not completed — Cycle cancellation | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMH Group | AFC Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [34 to 38] | 35 [33 to 37] | 35 [34 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 100 | 100 | 200
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Having Desired Ovarian Response
Description: Percentage of subjects with number of oocytes retrieved being between 6 and14
Time Frame: One single time point, i.e. at the time of oocyte retrieval
Population: Intention-to-treat basis. Those not proceeding with ovarian stimulation or oocyte retrieval were regarded as not having desired ovarian response
Measure: Count of Participants; unit: Participants
Arm/Group | AMH Group | AFC Group
Number analyzed (Participants) | 100 | 100
Participants | 49 | 54
Statistical Analysis 1: Comparison: AMH Group vs AFC Group; Test type: Superiority; p = 0.479, Chi-squared

2. Secondary Outcome: Percentage of Subjects Requiring Step-up or Step-down of Gonadotrophin Dose Upon First Ultrasound Tracking
Description: The dose of gonadotrophin will be adjusted according to the ovarian response: if 5 or less follicles growing beyond 10 mm --> step up if more than 15 follicles growing beyond 10 mm --> step down
Time Frame: 8th day of ovarian stimulation
Population: Intention-to-treat analysis. Two subjects in the AFC group did not proceed with treatment and were regarded as not requiring dosage adjustment.
Measure: Count of Participants; unit: Participants
Arm/Group | AMH Group | AFC Group
Number analyzed (Participants) | 100 | 100
Participants | 44 | 36
Statistical Analysis 1: Comparison: AMH Group vs AFC Group; Test type: Superiority; p = 0.002, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | AMH Group | AFC Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT02739269/Prot_SAP_000.pdf